CLINICAL TRIAL: NCT01891123
Title: An Open-label Randomized Clinical Trial to Compare the Toxicities and Efficacy of Pharmacokinetically-guided and BSA Fixed Dosing Strategy of Docetaxel and Paclitaxel in Chinese Non-small Cell Lung Cancer, Nasopharyngeal Carcinoma, and Breast Cancer Patients.
Brief Title: Explore the Individual Treatment of Docetaxel and Paclitaxel in NSCLC, NPC and BRC by PK-guided Dosing Strategy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li Zhang, Profressor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DT0508
Record Dates: First submitted 2013-06-18; First posted 2013-07-02 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Non-small Cell Lung Cancer; Breast Cancer; Nasal Cancer
Keywords: Non-small Cell Lung Cancer; Breast cancer; plasma drug concentration; Nasopharygeal carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Breast Neoplasms; Nose Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- body surface area (Placebo Comparator): patients receive fixed dose of PTX or DOC based on body surface area every cycle, PTX 175mg/m2, DOC 75mg/m2. Patients should finish up to 6 cycles chemotherapy
  Interventions: Drug: PTX 175mg/m2, DOC 75mg/m2
- Detection Kit (Active Comparator): PTX 175mg/m2, DOC 75mg/m2 at first cycle. the dose of PTX or DOC will adjust based on the pharmacokinetic results of previous cycle. A optimal target of PTX(TC>0.05) and DOC(AUC) have been set from published PK model with an established limited sampling strategy
  Interventions: Device: PK guided arm

INTERVENTIONS:
Device: PK guided arm — the dose of PTX or DOC will adjust based on the plasma drug concentration of previous cycle
  Other Names: pharmacokinetic guided dosing stratety
  Arms: Detection Kit
Drug: PTX 175mg/m2, DOC 75mg/m2 — patients receive PTX or DOC dose based on body surface area every cycle, PTX 175mg/m2, DOC 75mg/m2
  Arms: body surface area

SUMMARY:
As cytotoxic agents, DTX and PTX have a narrow therapeutic window. BSA dosing leads to great inter-individual PK variability, which is a major contributor for severe toxicity, especially in East-Asian populations. DTX exposures measured by area under plasma concentration-time curve (AUC), PTX exposures measured by the time above a plasma concentration of 0.05 µmol/L (TC>0.05), are the most biologic effects associated PK parameters for DTX and PTX, respectively, which could positively predict related toxicities such as neutropenia, peripheral neuropathy, etc. So, we conducted a randomized clinical trial to compare the effect on related toxicities and efficacy of PK-guided dosing strategy and BSA dosing strategy.

DETAILED DESCRIPTION:
3 populations were included: advanced NSCLC patients receive a single-agent docetaxel regimen palliative chemotherapy without restriction of lines; NPC patients receive paclitaxel and carboplatin doublet regimen whether as induction chemotherapy for local advanced patients or palliative chemotherapy for metastatic patients; BRC patients receive a single-agent docetaxel regimen after 4 cycles of adriamycin and cyclophosphamide for adjuvant chemotherapy. Patients are randomly assigned into the BSA-based dosing group and pharmacokinetically-guided dosing group. In the BSA-based dosing group, NPC patients receive paclitaxel (175mg/m2) and carboplatin (AUC=5) treatment, NSCLC and BRC patients receive docetaxel (75mg/m2) treatment, 3-weekly and for up to 6 cycles. BSA group and PK-guided group are with a same starting dose. DTX exposure (AUC) and PTX exposure (TC>0.05) are calculated from a published PK model with an established limited sampling strategy. Dose of subsequent cycles of PK-guided group patients is calculated base on the previous cycle PK results, according to optimal target algorithm. The optimal target for DTX exposure is 2.5 - 3.7 µg•h/mL. Dose reductions were permitted in both arms according to instructions. The study had a power of 80% to detect a 23% reduction of grade >3 neutropenia with PK-guided arm for DTX sub-study in NSCLC. A sample size of 100 NSCLC patients was estimated by using Fisher's exact test to provide a 5% two-sided alpha significance level to observe a decrease in the hematological toxicity with a power of 0.8. This is based on the reported toxicity rates of 85% with dose of 75mg/m2 and 63% with 60mg/m2. Objective response rate is evaluated by imaging examination (CT or MR scan) every 2 cycles. Toxicities are evaluated by patients' diary for toxicity reports and physician's evaluation at day 10 and day 21 at every cycle. Blood samples are collected every cycle. And survival information is collected by clinic and telephone follow-up. Research Hypothesis: 1. The concentrations variability dosed by BSA, and the limitation of BSA- and MTD-based dosing. 2. Verify that paclitaxel TC>0.05 and docetaxel AUC are the most relevant predictor of related toxicities and clinical outcomes. 3. Verify the feasibility of dosing algorithm based on paclitaxel TC>0.05 and docetaxel AUC, quantify its effect on both reducing toxicity and improving Effectiveness. 4. The effect of using dose modification and administration of G-CSF based on toxicity determined by paclitaxel TC>0.05 and docetaxel AUC measurement. 5. Prove the ability of PK-guided dosing strategy in reducing DTX and PTX related hematologic and non-hematologic toxicities, and the effect on treatment efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed by pathology for advanced non small cell lung cancer, suitable for paclitaxel or docetaxel chemotherapy (clinical stage IV according to 2009 IASLC staging or recurrent NSCLC; receiving palliative chemotherapy independent of lines)
* ECOG PS score: 0 to 2 points
* Survival is expected to more than 3 month
* Bone marrow reserve function is good, the function of organs (liver and kidney) is good, can satisfy the conditions of implementation chemotherapy.
* Sign the informed consent form
* Compliance is good, can be followed up, willing to comply with the requirements of the study

Exclusion Criteria:

* Physical status score (ECOG) greater than 2
* organic disease；Severely active infection；Organ transplantation immune therapy；Can't complete with in four to six cycles of chemotherapy
* Bone marrow, liver and kidney dysfunction, clinical doctors identify intolerance to chemotherapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2013-06; Primary Completion 2016-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Toxicities rate | 3 weeks, 6 weeks, 9 weeks, 12 weeks, 15 weeks, 18weeks
  assess the toxicities rate and severity according to CTCAE v4.03, record the toxicities incident and grades from the first cycle to last cycle until the toxicities relieve or stabilize.

SECONDARY OUTCOMES:
Object response rate | up to 18 weeks
  assess the ORR according to RECIST v1.1, An imaging examination should be performed in 4weeks before treatment initiation, and patients are going to receive (CT or MR scan) every 2 cycles during the treatment, the methods should be identical with baseline.
Survival Effectiveness | 36 months
  after treatment discontinuation, PFS is recorded by imaging examination every 2 cycles (8 weeks) until tumor progression, other anti-cancer treatment start, trial ends or death. OS is recorded by clinic follow-up or telephone follow-up until death.

OTHER OUTCOMES:
the quality of life of patients | 3 weeks, 6 weeks, 9 weeks, 12 weeks, 15 weeks, 18weeks

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, Principal Investigator — Sun Yat-sen University; Shu Sen Wang, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Cao SM, Simons MJ, Qian CN. The prevalence and prevention of nasopharyngeal carcinoma in China. Chin J Cancer. 2011 Feb;30(2):114-9. doi: 10.5732/cjc.010.10377. PMID 21272443
- [Background] Chan AT, Ma BB, Lo YM, Leung SF, Kwan WH, Hui EP, Mok TS, Kam M, Chan LS, Chiu SK, Yu KH, Cheung KY, Lai K, Lai M, Mo F, Yeo W, King A, Johnson PJ, Teo PM, Zee B. Phase II study of neoadjuvant carboplatin and paclitaxel followed by radiotherapy and concurrent cisplatin in patients with locoregionally advanced nasopharyngeal carcinoma: therapeutic monitoring with plasma Epstein-Barr virus DNA. J Clin Oncol. 2004 Aug 1;22(15):3053-60. doi: 10.1200/JCO.2004.05.178. PMID 15284255
- [Background] Miyaushiro S, Kitanaka A, Kubuki Y, Hidaka T, Shide K, Kameda T, Sekine M, Kamiunten A, Umekita Y, Kawabata T, Ishiguro Y, Shimoda K. Nasopharyngeal carcinoma with bone marrow metastasis: positive response to weekly paclitaxel chemotherapy. Intern Med. 2015;54(11):1455-9. doi: 10.2169/internalmedicine.54.3917. Epub 2015 Jun 1. PMID 26028007
- [Background] Ciuleanu TE, Fountzilas G, Ciuleanu E, Plataniotis M, Todor N, Ghilezan N. Paclitaxel and carboplatin in relapsed or metastatic nasopharyngeal carcinoma: a multicenter phase II study. J BUON. 2004 Apr-Jun;9(2):161-5. PMID 17415808
- [Background] Tan EH, Khoo KS, Wee J, Fong KW, Lee KS, Lee KM, Chua ET, Tan T, Khoo-Tan HS, Yang TL, Au E, Tao M, Ong YK, Chua EJ. Phase II trial of a paclitaxel and carboplatin combination in Asian patients with metastatic nasopharyngeal carcinoma. Ann Oncol. 1999 Feb;10(2):235-7. doi: 10.1023/a:1008390929826. PMID 10093695
- [Background] Undevia SD, Gomez-Abuin G, Ratain MJ. Pharmacokinetic variability of anticancer agents. Nat Rev Cancer. 2005 Jun;5(6):447-58. doi: 10.1038/nrc1629. PMID 15928675
- [Background] Baker SD, Verweij J, Rowinsky EK, Donehower RC, Schellens JH, Grochow LB, Sparreboom A. Role of body surface area in dosing of investigational anticancer agents in adults, 1991-2001. J Natl Cancer Inst. 2002 Dec 18;94(24):1883-8. doi: 10.1093/jnci/94.24.1883. PMID 12488482
- [Background] Engels FK, Loos WJ, van der Bol JM, de Bruijn P, Mathijssen RH, Verweij J, Mathot RA. Therapeutic drug monitoring for the individualization of docetaxel dosing: a randomized pharmacokinetic study. Clin Cancer Res. 2011 Jan 15;17(2):353-62. doi: 10.1158/1078-0432.CCR-10-1636. Epub 2011 Jan 11. PMID 21224369
- [Background] Rudek MA, Sparreboom A, Garrett-Mayer ES, Armstrong DK, Wolff AC, Verweij J, Baker SD. Factors affecting pharmacokinetic variability following doxorubicin and docetaxel-based therapy. Eur J Cancer. 2004 May;40(8):1170-8. doi: 10.1016/j.ejca.2003.12.026. PMID 15110880
- [Background] Bruno R, Hille D, Riva A, Vivier N, ten Bokkel Huinnink WW, van Oosterom AT, Kaye SB, Verweij J, Fossella FV, Valero V, Rigas JR, Seidman AD, Chevallier B, Fumoleau P, Burris HA, Ravdin PM, Sheiner LB. Population pharmacokinetics/pharmacodynamics of docetaxel in phase II studies in patients with cancer. J Clin Oncol. 1998 Jan;16(1):187-96. doi: 10.1200/JCO.1998.16.1.187. PMID 9440742
- [Background] Rosing H, Lustig V, van Warmerdam LJ, Huizing MT, ten Bokkel Huinink WW, Schellens JH, Rodenhuis S, Bult A, Beijnen JH. Pharmacokinetics and metabolism of docetaxel administered as a 1-h intravenous infusion. Cancer Chemother Pharmacol. 2000;45(3):213-8. doi: 10.1007/s002800050032. PMID 10663639
- [Background] Bruno R, Vivier N, Veyrat-Follet C, Montay G, Rhodes GR. Population pharmacokinetics and pharmacokinetic-pharmacodynamic relationships for docetaxel. Invest New Drugs. 2001 May;19(2):163-9. doi: 10.1023/a:1010687017717. PMID 11392450
- [Background] Baker SD, Li J, ten Tije AJ, Figg WD, Graveland W, Verweij J, Sparreboom A. Relationship of systemic exposure to unbound docetaxel and neutropenia. Clin Pharmacol Ther. 2005 Jan;77(1):43-53. doi: 10.1016/j.clpt.2004.09.005. PMID 15637530
- [Background] Extra JM, Rousseau F, Bruno R, Clavel M, Le Bail N, Marty M. Phase I and pharmacokinetic study of Taxotere (RP 56976; NSC 628503) given as a short intravenous infusion. Cancer Res. 1993 Mar 1;53(5):1037-42. PMID 8094996
- [Background] Minami H, Kawada K, Sasaki Y, Igarashi T, Saeki T, Tahara M, Itoh K, Fujii H. Pharmacokinetics and pharmacodynamics of protein-unbound docetaxel in cancer patients. Cancer Sci. 2006 Mar;97(3):235-41. doi: 10.1111/j.1349-7006.2006.00166.x. PMID 16542221
- [Background] Minami H, Ohe Y, Niho S, Goto K, Ohmatsu H, Kubota K, Kakinuma R, Nishiwaki Y, Nokihara H, Sekine I, Saijo N, Hanada K, Ogata H. Comparison of pharmacokinetics and pharmacodynamics of docetaxel and Cisplatin in elderly and non-elderly patients: why is toxicity increased in elderly patients? J Clin Oncol. 2004 Jul 15;22(14):2901-8. doi: 10.1200/JCO.2004.10.163. PMID 15254059
- [Background] Minami H, Kawada K, Sasaki Y, Tahara M, Igarashi T, Itoh K, Fujii H, Saeki T, Ozawa K, Sato H. Population pharmacokinetics of docetaxel in patients with hepatic dysfunction treated in an oncology practice. Cancer Sci. 2009 Jan;100(1):144-9. doi: 10.1111/j.1349-7006.2009.00992.x. Epub 2008 Oct 30. PMID 19018756
- [Background] Ozawa K, Minami H, Sato H. Logistic regression analysis for febrile neutropenia (FN) induced by docetaxel in Japanese cancer patients. Cancer Chemother Pharmacol. 2008 Aug;62(3):551-7. doi: 10.1007/s00280-007-0648-8. Epub 2007 Dec 7. PMID 18064462
- [Background] Ozawa K, Minami H, Sato H. Clinical trial simulations for dosage optimization of docetaxel in patients with liver dysfunction, based on a log-binominal regression for febrile neutropenia. Yakugaku Zasshi. 2009 Jun;129(6):749-57. doi: 10.1248/yakushi.129.749. PMID 19483418
- [Background] Ghersi D, Wilcken N, Simes RJ. A systematic review of taxane-containing regimens for metastatic breast cancer. Br J Cancer. 2005 Aug 8;93(3):293-301. doi: 10.1038/sj.bjc.6602680. PMID 16052223
- [Background] Henderson IC, Berry DA, Demetri GD, Cirrincione CT, Goldstein LJ, Martino S, Ingle JN, Cooper MR, Hayes DF, Tkaczuk KH, Fleming G, Holland JF, Duggan DB, Carpenter JT, Frei E 3rd, Schilsky RL, Wood WC, Muss HB, Norton L. Improved outcomes from adding sequential Paclitaxel but not from escalating Doxorubicin dose in an adjuvant chemotherapy regimen for patients with node-positive primary breast cancer. J Clin Oncol. 2003 Mar 15;21(6):976-83. doi: 10.1200/JCO.2003.02.063. PMID 12637460
- [Background] Martin M, Rodriguez-Lescure A, Ruiz A, Alba E, Calvo L, Ruiz-Borrego M, Munarriz B, Rodriguez CA, Crespo C, de Alava E, Lopez Garcia-Asenjo JA, Guitian MD, Almenar S, Gonzalez-Palacios JF, Vera F, Palacios J, Ramos M, Gracia Marco JM, Lluch A, Alvarez I, Segui MA, Mayordomo JI, Anton A, Baena JM, Plazaola A, Modolell A, Pelegri A, Mel JR, Aranda E, Adrover E, Alvarez JV, Garcia Puche JL, Sanchez-Rovira P, Gonzalez S, Lopez-Vega JM; GEICAM 9906 Study Investigators. Randomized phase 3 trial of fluorouracil, epirubicin, and cyclophosphamide alone or followed by Paclitaxel for early breast cancer. J Natl Cancer Inst. 2008 Jun 4;100(11):805-14. doi: 10.1093/jnci/djn151. Epub 2008 May 27. PMID 18505968
- [Background] Bear HD, Anderson S, Smith RE, Geyer CE Jr, Mamounas EP, Fisher B, Brown AM, Robidoux A, Margolese R, Kahlenberg MS, Paik S, Soran A, Wickerham DL, Wolmark N. Sequential preoperative or postoperative docetaxel added to preoperative doxorubicin plus cyclophosphamide for operable breast cancer:National Surgical Adjuvant Breast and Bowel Project Protocol B-27. J Clin Oncol. 2006 May 1;24(13):2019-27. doi: 10.1200/JCO.2005.04.1665. Epub 2006 Apr 10. PMID 16606972
- [Background] Jones SE, Savin MA, Holmes FA, O'Shaughnessy JA, Blum JL, Vukelja S, McIntyre KJ, Pippen JE, Bordelon JH, Kirby R, Sandbach J, Hyman WJ, Khandelwal P, Negron AG, Richards DA, Anthony SP, Mennel RG, Boehm KA, Meyer WG, Asmar L. Phase III trial comparing doxorubicin plus cyclophosphamide with docetaxel plus cyclophosphamide as adjuvant therapy for operable breast cancer. J Clin Oncol. 2006 Dec 1;24(34):5381-7. doi: 10.1200/JCO.2006.06.5391. PMID 17135639
- [Background] O'Shaughnessy J, Miles D, Vukelja S, Moiseyenko V, Ayoub JP, Cervantes G, Fumoleau P, Jones S, Lui WY, Mauriac L, Twelves C, Van Hazel G, Verma S, Leonard R. Superior survival with capecitabine plus docetaxel combination therapy in anthracycline-pretreated patients with advanced breast cancer: phase III trial results. J Clin Oncol. 2002 Jun 15;20(12):2812-23. doi: 10.1200/JCO.2002.09.002. PMID 12065558
- [Background] Sparano JA, Wang M, Martino S, Jones V, Perez EA, Saphner T, Wolff AC, Sledge GW Jr, Wood WC, Davidson NE. Weekly paclitaxel in the adjuvant treatment of breast cancer. N Engl J Med. 2008 Apr 17;358(16):1663-71. doi: 10.1056/NEJMoa0707056. PMID 18420499
- [Background] Milano G, Etienne MC, Renee N, Thyss A, Schneider M, Ramaioli A, Demard F. Relationship between fluorouracil systemic exposure and tumor response and patient survival. J Clin Oncol. 1994 Jun;12(6):1291-5. doi: 10.1200/JCO.1994.12.6.1291. PMID 8201391
- [Background] Gambacorti-Passerini C, Zucchetti M, Russo D, Frapolli R, Verga M, Bungaro S, Tornaghi L, Rossi F, Pioltelli P, Pogliani E, Alberti D, Corneo G, D'Incalci M. Alpha1 acid glycoprotein binds to imatinib (STI571) and substantially alters its pharmacokinetics in chronic myeloid leukemia patients. Clin Cancer Res. 2003 Feb;9(2):625-32. PMID 12576428
- [Background] Alexandre J, Rey E, Girre V, Grabar S, Tran A, Montheil V, Rabillon F, Dieras V, Jullien V, Herait P, Pons G, Treluyer JM, Goldwasser F. Relationship between cytochrome 3A activity, inflammatory status and the risk of docetaxel-induced febrile neutropenia: a prospective study. Ann Oncol. 2007 Jan;18(1):168-172. doi: 10.1093/annonc/mdl321. Epub 2006 Oct 23. PMID 17060489
- [Background] Huizing MT, Keung AC, Rosing H, van der Kuij V, ten Bokkel Huinink WW, Mandjes IM, Dubbelman AC, Pinedo HM, Beijnen JH. Pharmacokinetics of paclitaxel and metabolites in a randomized comparative study in platinum-pretreated ovarian cancer patients. J Clin Oncol. 1993 Nov;11(11):2127-35. doi: 10.1200/JCO.1993.11.11.2127. PMID 7901342
- [Background] Sarosy G, Reed E. Taxol dose intensification and its clinical implications. J Natl Med Assoc. 1993 Jun;85(6):427-31. PMID 8103561
- [Background] Huizing MT, Giaccone G, van Warmerdam LJ, Rosing H, Bakker PJ, Vermorken JB, Postmus PE, van Zandwijk N, Koolen MG, ten Bokkel Huinink WW, van der Vijgh WJ, Bierhorst FJ, Lai A, Dalesio O, Pinedo HM, Veenhof CH, Beijnen JH. Pharmacokinetics of paclitaxel and carboplatin in a dose-escalating and dose-sequencing study in patients with non-small-cell lung cancer. The European Cancer Centre. J Clin Oncol. 1997 Jan;15(1):317-29. doi: 10.1200/JCO.1997.15.1.317. PMID 8996159
- [Background] Joerger M, Huitema AD, Richel DJ, Dittrich C, Pavlidis N, Briasoulis E, Vermorken JB, Strocchi E, Martoni A, Sorio R, Sleeboom HP, Izquierdo MA, Jodrell DI, Calvert H, Boddy AV, Hollema H, Fety R, Van der Vijgh WJ, Hempel G, Chatelut E, Karlsson M, Wilkins J, Tranchand B, Schrijvers AH, Twelves C, Beijnen JH, Schellens JH. Population pharmacokinetics and pharmacodynamics of paclitaxel and carboplatin in ovarian cancer patients: a study by the European organization for research and treatment of cancer-pharmacology and molecular mechanisms group and new drug development group. Clin Cancer Res. 2007 Nov 1;13(21):6410-8. doi: 10.1158/1078-0432.CCR-07-0064. PMID 17975154
- [Background] Miller AA, Rosner GL, Egorin MJ, Hollis D, Lichtman SM, Ratain MJ. Prospective evaluation of body surface area as a determinant of paclitaxel pharmacokinetics and pharmacodynamics in women with solid tumors: Cancer and Leukemia Group B Study 9763. Clin Cancer Res. 2004 Dec 15;10(24):8325-31. doi: 10.1158/1078-0432.CCR-04-1078. PMID 15623609
- [Background] Ohtsu T, Sasaki Y, Tamura T, Miyata Y, Nakanomyo H, Nishiwaki Y, Saijo N. Clinical pharmacokinetics and pharmacodynamics of paclitaxel: a 3-hour infusion versus a 24-hour infusion. Clin Cancer Res. 1995 Jun;1(6):599-606. PMID 9816021
- [Background] Gianni L, Kearns CM, Giani A, Capri G, Vigano L, Lacatelli A, Bonadonna G, Egorin MJ. Nonlinear pharmacokinetics and metabolism of paclitaxel and its pharmacokinetic/pharmacodynamic relationships in humans. J Clin Oncol. 1995 Jan;13(1):180-90. doi: 10.1200/JCO.1995.13.1.180. PMID 7799018
- [Background] Jiko M, Yano I, Sato E, Takahashi K, Motohashi H, Masuda S, Okuda M, Ito N, Nakamura E, Segawa T, Kamoto T, Ogawa O, Inui K. Pharmacokinetics and pharmacodynamics of paclitaxel with carboplatin or gemcitabine, and effects of CYP3A5 and MDR1 polymorphisms in patients with urogenital cancers. Int J Clin Oncol. 2007 Aug;12(4):284-90. doi: 10.1007/s10147-007-0681-y. Epub 2007 Aug 20. PMID 17701008
- [Background] Mielke S, Sparreboom A, Steinberg SM, Gelderblom H, Unger C, Behringer D, Mross K. Association of Paclitaxel pharmacokinetics with the development of peripheral neuropathy in patients with advanced cancer. Clin Cancer Res. 2005 Jul 1;11(13):4843-50. doi: 10.1158/1078-0432.CCR-05-0298. PMID 16000582
- [Background] Joerger M, Huitema AD, van den Bongard DH, Schellens JH, Beijnen JH. Quantitative effect of gender, age, liver function, and body size on the population pharmacokinetics of Paclitaxel in patients with solid tumors. Clin Cancer Res. 2006 Apr 1;12(7 Pt 1):2150-7. doi: 10.1158/1078-0432.CCR-05-2069. PMID 16609028